CLINICAL TRIAL: NCT02344836
Title: Refining and Pilot Testing Social Networks for Encouraging Healthy Behaviors: The Social Pounds Off Digitally (Social POD) Study
Brief Title: The Social Pounds Off Digitally (Social POD) Study
Acronym: SocialPOD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Brie Turner-McGrievy, Assistant professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00034960
Record Dates: First submitted 2015-01-16; First posted 2015-01-26 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Theory-based podcast (Active Comparator): Receive a 3-month weight loss intervention delivered via theory-based podcast (TBP) plus self-monitoring using a commercially-available calorie and weight tracking app (current most popular diet self-monitoring method).
  Intervention: podcast + mobile diet app
  Interventions: Behavioral: Podcast + mobile diet app
- Theory-based podcast + Social POD (Experimental): Receive a 3-month weight loss intervention delivered via Theory-based Podcast (TBP) plus self-monitoring and social support/incentive points for participating with the Social POD app (TBP+Social POD).
  Intervention: podcast + theory-based mobile diet app
  Interventions: Behavioral: Podcast + theory-based mobile diet app

INTERVENTIONS:
Behavioral: Podcast + mobile diet app — Use of a mobile app to track behaviors related to weight loss as well as receive study-related weight loss information via podcast.
  Arms: Theory-based podcast
Behavioral: Podcast + theory-based mobile diet app — Use of a theory-based mobile app to track behaviors related to weight loss as well as receive study-related weight loss information via podcast.
  Arms: Theory-based podcast + Social POD

SUMMARY:
Smartphones have the capability to monitor health-related behaviors (exercise, diet, etc.) and provide social support which has the potential to play a powerful role in health promotion. The objective of this study is to refine and pilot test the Social POD app for personalized health monitoring and interaction founded on a combination of social networks, recommender systems, motivational research, and health behavior theory. The aim of our proposed project is to conduct a 3-month pilot RCT among overweight and obese adults (N=150) comparing a theory-based podcast (TBP) plus self-monitoring using a commercially-available calorie and weight tracking app (current most popular diet self-monitoring method) versus TBP plus self-monitoring and social support/incentive points for participating with the Social POD app (TBP+Social POD).

DETAILED DESCRIPTION:
Objectives and Significance. Smartphones have the capability to monitor health-related behaviors (exercise, diet, etc.) and provide social support which has the potential to play a powerful role in health promotion. The objective of this study is to refine and pilot test the Social POD app for personalized health monitoring and interaction founded on a combination of social networks, recommender systems, motivational research, and health behavior theory. Currently, we are recruiting for usability testing among obese and overweight (BMI >25 kg/m2) adults (n=20) with our basic Social POD app. Our proposed project, which seeks to supplement our current line of research investigating mHealth interventions for overweight and obese adults, has two aims:

Aim 1: Refine our intelligent social agent mobile app (Social POD) based on results from our usability testing and develop new components (i.e., incentive system) for use in a 3-month randomized controlled pilot trial (RCT).

Aim 2: Conduct a 3-month pilot RCT among overweight and obese adults (N=150) comparing a theory-based podcast (TBP) plus self-monitoring using a commercially-available calorie and weight tracking app (current most popular diet self-monitoring method)9 versus TBP plus self-monitoring and social support/incentive points for participating with the Social POD app (TBP+Social POD).

Once the final intervention is developed through Aim 1 including the incentive system, we will recruit 150 overweight adult Android smartphone owners (BMI 25-49.9 kg/m2; age 18-65; >30% AA) to participate in a 3-month pilot of our enhanced intervention. Detecting differences in weight among the two groups is our primary research goal.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese (Body Mass Index between 25 and 49.9 kg/m2)
* Own and Android phone or tablet

Exclusion Criteria:

* are currently pregnant
* are younger than 18 or older than 65 years of age
* are unable to attend 3 meetings at the University of South Carolina
* don't have access to the Internet and a computer
* don't have access to a scale for self-monitoring weight
* aren't willing to be randomized to one of the two groups
* have a psychiatric disease, drug or alcohol dependency, or uncontrolled thyroid condition
* have a major health condition, such as heart conditions, diabetes, and past incidence of stroke
* have an eating disorder
* currently participating in a weight loss program or taking weight loss medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Weight loss | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Hales S, Turner-McGrievy GM, Wilcox S, Davis RE, Fahim A, Huhns M, Valafar H. Trading pounds for points: Engagement and weight loss in a mobile health intervention. Digit Health. 2017 Apr 24;3:2055207617702252. doi: 10.1177/2055207617702252. eCollection 2017 Jan-Dec. PMID 29942590
- [Derived] Hales S, Turner-McGrievy GM, Wilcox S, Fahim A, Davis RE, Huhns M, Valafar H. Social networks for improving healthy weight loss behaviors for overweight and obese adults: A randomized clinical trial of the social pounds off digitally (Social POD) mobile app. Int J Med Inform. 2016 Oct;94:81-90. doi: 10.1016/j.ijmedinf.2016.07.003. Epub 2016 Jul 2. PMID 27573315